CLINICAL TRIAL: NCT04163055
Title: The F.L.I.G.H.T. (Fluorescence Image-Guided Healing Trial) for Diabetic Foot Ulcers: A Phase IV Trial
Brief Title: Fluorescence Image-Guided Healing Trial
Acronym: FLIGHT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-6034
Record Dates: First submitted 2019-11-07; First posted 2019-11-14 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Diabetic Foot Ulcer
Keywords: Diabetes; Foot Ulcer; Non-healing wound; Targeted debridement
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus; Foot Ulcer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standard of Care (No Intervention): Wounds will be assessed using the Clinical Signs and Symptoms Checklist (CSSC). After initial assessment, a white-light (WL) photo will be taken of the wound. The wound bed will be prepared as indicated by clinical staff based on standard of care (SoC), including irrigation and debridement. A second WL image will be taken and a swab/biopsy will be obtained from the wound. Wounds will be dressed based on SoC.
- Autofluorescence guided Standard of Care (Experimental): Wounds will be assessed by autofluorescence (AF)-guided SoC. A baseline WL and AF photo will be taken of the wound. AF images will guide SoC including targeted debridement of areas of bacterial growth (AF+) and targeted sampling in areas of residual bacterial growth post-debridement. If no bacterial AF is detected, sample will be obtained from the wound center by curettage technique. If AF is detected, AF-guided debridement will be repeated and additional images will be obtained until 1) no AF is detected or 2) further debridement is not medically advised. After wound bed preparation, a second set of WL and AF images will be taken. Wounds will be dressed as per SoC. At all visits, samples will be sent for microbiology analysis. At 6- and 12-week visits (or any other scheduled visits in between), microbiology reports will be shared with clinicians if they were not collected outside of SoC.
  Interventions: Device: Moleculight i:X

INTERVENTIONS:
Device: Moleculight i:X — This device is used to visualize the bacteria in the wound. Patients do not need consume any contrast agent prior to imaging. The device does not come in contact with the wound.
  Arms: Autofluorescence guided Standard of Care

SUMMARY:
Lower extremity complications such as chronic diabetic foot ulcers (DFUs) are a major risk for Type I/II diabetes patients. Minor injuries that would normally heal without consequence in non-diabetic individuals are at greater risk of bacterial infection and progression to non healing (chronic) wound status in diabetics, largely due to a loss of sensation in limbs (neuropathy) and decreased blood flow (vascular disease). If not treated efficiently and effectively, DFUs can have serious complications e.g. amputation, sepsis and death. The investigators propose to address this significant unmet clinical need using a novel commercial handheld fluorescence imaging product called the MolecuLight i:X (MolecuLight Inc.) which images clinically-significant wound bacteria without contrast agents or patient contact. Evidence in animal models of chronic wounds and multiple published clinical trials (mainly DFUs) have shown significant clinical potential for fluorescence imaging to detect potentially harmful bacteria in wounds otherwise invisible to doctors. The investigators have shown that clinicians can easily, objectively and more accurately determine the likelihood of bacterial infection than the standard of care. Moreover, published clinical evidence has shown fluorescence imaging enables more accurate microbial wound sampling and guides more targeted debridement of wounds to reduce bacteria levels. Our pilot data also show that when used like this, the i:X device accelerates DFU wound healing, compared with current methods. Thus, the investigators propose to expand the current pilot studies through a statistically-powered 3 y randomized controlled trial to test the therapeutic benefit of fluorescence-guided treatment for DFUs in a larger group of patients. A successful trial could help reduce DFU healing times compared with standard practice (using a new Canadian product) and improve patient quality of life, reduce amputation risk and alleviate health care costs for diabetes complications in Canada and beyond.

DETAILED DESCRIPTION:
Wound care is a major clinical challenge and presents an enormous burden to health care worldwide. Wounds Canada describes chronic wounds as "a Canadian healthcare crisis." According to Wounds Canada and Diabetes Canada, approximately 15% of the 2.3 million diabetic Canadians will develop a diabetic foot ulcer (DFU) and every 30 seconds someone in the world loses a toe or limb to diabetes. Diabetics are about 23x more likely to be hospitalized for amputations, approximately 85% of which are due to a previous DFU. Delayed wound healing has been linked to a variety of factors including infection, which disrupts key biological changes at the tissue and cellular level that are associated with the wound healing process. Standard of care (SoC) of DFU infections involves visual inspection of the wound under white light (WL) and identification of common signs of infection using the Clinical Signs and Symptoms Checklist. However, SoC is limited by inconsistent guidelines and subjective assessment. In addition, visual inspection and WL-guided sampling are inaccurate and currently, no point-of-care technologies exist to assist the unaided eye. In response to this gap, Dr. DaCosta (PI) and colleagues at University Health Network developed a handheld fluorescence imaging platform (MolecuLight i:X) that detects bacterial autofluorescence in wounds in real-time, at the point-of-care, and without the use of exogenous contrast agents. The investigators propose a 3-year randomized control trial to test the therapeutic benefit of AF-image guided intervention on DFU management using the i:X. The research questions are Q1). Does AF-guided diagnosis and wound bed preparation improve wound healing in DFUs relative to SoC alone? Q2). Does AF-guided intervention decrease the bioburden in DFUs relative to SoC alone? Q3). Does AF-guided intervention improve patient quality of life relative to SoC alone? Q4). Is AF-guided intervention associated with reduced treatment cost? Primary objective: is to determine if AF-guided diagnosis and wound bed preparation improve wound healing in DFUs compared to SoC alone. To measure this, the investigators will compare between study arms i) the frequency of complete wound healing (CWH) at 12 weeks; ii) the frequency of partial wound healing (PWH) at 6 and 12 weeks, CWH at 6 weeks, and mean time-to-CWH (days); iii) the reduction in wound size at 12 weeks; and iv) the rate of wound healing over 12 weeks. Secondary objective: is to determine if AF-guided intervention decreases the bioburden in DFUs compared to SoC alone by evaluating bacterial diversity and measuring bacteria load at specified regular intervals over 12 weeks. Tertiary objective: is to determine if AF-guided intervention is associated with improved quality of life (QoL) and with reduced treatment costs, which will be measured by using patient questionnaires and the Canadian Institute for Health Information database.

If successful, this Randomized Control Trial (RCT) will demonstrate that AF image-guided wound care improves time to CWH or PWH among Ontarians with DFUs by increasing wound healing rates and reducing bioburden. If our technology can improve CWH by our target of >= 16% (absolute), an additional 55,000 Canadians could reach CWH by 12 weeks, resulting in reduced wound care costs and improved QoL. The average cost of treating a DFU is $5000-8000/patient. Improving the number of patients that achieve CWH by >= 16% will substantially reduce costs associated with treating DFUs in Canada. The results of this study may inform health policy decisions and recommendations for changes to current SoC DFU practice guidelines. Health economic and QoL comparison of AF-guided wound care vs SoC in the proposed RCT will help define the overall value proposition of the new approach. If the investigators fail to demonstrate improved wound healing rates, this will also be of value to physicians, patients and the Canadian health care system. Knowing not to further pursue this line of research is important in an era of limited funding.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with type I or II diabetes
2. Presents with one or more chronic or acute DFUs of known or unknown infection status
3. Presents with a DFU with surface area that has reduced <25% in the last 4 weeks
4. Braden Score ≥13-14 (Moderate Risk)
5. Toe-Brachial Index > 0.5 (Mild-Normal)

Exclusion Criteria:

1. Wounds < 1 cm in diameter
2. Current or past (within 1 month) treatment of DFU with antibiotics
3. Treatment with an investigational drug within 1 month of enrolment
4. Presents with chronic (>10mg/kg for >30 days) systemic corticoids before enrolment
5. Undergoing chemotherapy or is immunocompromised
6. Diagnosed with Charcot disease or ulcers from electrical, chemical or radiation burns
7. Presents with collagen vascular disease, ulcer malignancy, cellulitis, or chronic osteomyelitis (defined as a severe, persistent and sometimes incapacitating infection of bone and bone marrow).
8. Recombinant or autologous growth factors or skin/dermal substitutes within 30 days of enrollment
9. Enzymatic debridement
10. Acquired a limb-threatening infection which necessitates an amputation
11. InfectionHas a terminal illness
12. Inability to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
The rate of CWH of DFUs will be estimated as a proportion and compared between the two groups using a chi square test. The superiority of AF-guided intervention (Arm 2) will be established if the null hypothesis is rejected. | 12 weeks
  CWH is defined as 100% re-epithelialization, and will be recorded and validated by independent review. The % of patients achieving CWH will be evaluated at 6- and 12-wk and compared between study arms (time point based on previously published data regarding wound healing in DFUs). Time to CWH will also be recorded and compared between study arms. PWH is defined as a reduction in wound area (WA) of ≥50% relative to baseline, but not meeting criteria of CWH. The % of patients achieving PWH will be evaluated at 6 and 12-wk and compared between study arms. To validate CWH, images of wounds identified as having reached 100% re-epithelialization by the wound care clinician will be photographed under WL and sent for review by at least 2 independent blinded researchers.

SECONDARY OUTCOMES:
Rate of Wound Healing | 12 weeks
  The rate of PWH of DFUs at 6 and 12 weeks and CWH at 6 weeks will be estimated as a proportion and compared between the two groups using chi-square analysis
The percent reduction in wound area | 12 weeks
  Wound area reduction at 6 and 12 weeks will be estimated as an average percent wound area reduction relative to baseline and will be compared between the two groups using Student's t-test and linear regression (adjusting for risk factors related to change in wound area).
The bioburden of the wound identified and quantified | 12 weeks
  Clinical microbiology reports (from curettage samples) will be used to determine wound bioburden, defined as the diversity of species and semi-quantitative bacterial load.
To evaluate cost effectiveness and cost utility of the device on treatment | 12 weeks
  An economic analysis will be conducted to evaluate the cost-effectiveness and cost-utility of the i:X intervention relative to standard of care (SoC) for patients with diabetic foot ulcers.
Quality of Life improvement due to the device as assessed by EuroQol-5D-5L | 12 weeks
  The health outcome for the cost-effectiveness analysis will be the proportion of patients with complete wound healing at 12 weeks post initial intervention (same as the primary study end-point).The health outcome for the cost-utility analysis will be quality adjusted life years (QALYs). Quality of life will be measured throughout the trial using the EuroQoL Five Dimensions (EQ-5D-5L) instrument (Scale is between 0-100, with 100 being the best health you can imaging and 0 being the worst health you can imagine) .
Quality of Life improvement due to the device as assessed by Short Form -12 Health Questionnaire | 12 weeks
  The health outcome for the cost-effectiveness analysis will be the proportion of patients with complete wound healing at 12 weeks post initial intervention (same as the primary study end-point).The health outcome for the cost-utility analysis will be quality adjusted life years (QALYs). Quality of life will be measured throughout the trial using the Short Form -12 Health questionnaire instrument (On a scale of 1(all the time) - 6(none of the time) and 1(yes limited a lot) -3 (no not limited at all)).
Quality of Life improvement due to the device as assessed Diabetic Foot Ulcer Scale | 12 weeks
  The health outcome for the cost-effectiveness analysis will be the proportion of patients with complete wound healing at 12 weeks post initial intervention (same as the primary study end-point).The health outcome for the cost-utility analysis will be quality adjusted life years (QALYs). Quality of life will be measured throughout the trial using the Diabetic Foot Ulcer Scale instrument (The scale for this instrument is 1 to 5 with 1 being not likely to 5 being extremely likely).

IPD SHARING:
Plan to Share IPD: No